CLINICAL TRIAL: NCT00030407
Title: Evaluation Of Celecoxib In Combination With Weekly Docetaxel In Elderly (70 Years) Or Poor Performance Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Celecoxib and Docetaxel in Treating Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069163; P30CA022453 (NIH); WSU-C-2305 (Other: Barbara Ann Karmanos Cancer Institute); NCI-V01-1687
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Celecoxib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Celecoxib & Docetaxel (Experimental): Celecoxib: On day -7 of the first cycle, patients will start, Celecoxib 400 mg po bid daily, each dose to give with meals
  Docetaxel: On day 1, 8, and 15 of each cycle patients will receive: Docetaxel 36mg/m2 over 60 minutes, duration of each cycle will be 28 days.
  Interventions: Drug: Celecoxib; Drug: Docetaxel

INTERVENTIONS:
Drug: Celecoxib — On day -7 of the first cycle, patients will start, Celecoxib 400 mg po bid daily, each dose to give with meals
  Other Names: Celebrex; Celebra
Drug: Docetaxel — On day 1, 8, and 15 of each cycle patients will receive: Docetaxel 36mg/m2 over 60 minutes, duration of each cycle will be 28 days.
  Other Names: Taxotere®

SUMMARY:
RATIONALE: Celecoxib may slow the growth of cancer by stopping blood flow to the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy and celecoxib may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of celecoxib and docetaxel in treating patients who have non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy and feasibility of celecoxib combined with docetaxel as first-line therapy in elderly or poor performance status patients with advanced non-small cell lung cancer.
* Determine the response rate of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral celecoxib twice daily (beginning on day -7 of the first course) and docetaxel IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients who achieve a complete response (CR) receive 2 additional courses after CR. Patients who achieve stable disease (SD) or a partial response (PR) receive a minimum of 2 additional courses after SD or PR. At the discretion of the treating physician, patients then receive maintenance therapy comprising celecoxib only.

Patients who discontinue therapy for disease progression or unacceptable toxicity are followed for at least 6 months.

PROJECTED ACCRUAL: A total of 21-39 patients will be accrued for this study within 13-28 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-small cell lung cancer (NSCLC)

  * Stage IIIB with pleural effusion or stage IV disease
* Age 70 years and over with SWOG performance status 0-2 OR age 18 to 69 with SWOG performance status 2
* Measurable or evaluable disease
* No symptomatic or untreated brain or leptomeningeal metastases

  * Previously treated patients must be neurologically stable for 4 weeks after completion of appropriate therapy

PATIENT CHARACTERISTICS:

Age:

* See Disease Characteristics
* 18 and over

Performance status:

* See Disease Characteristics
* SWOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* AST/ALT no greater than ULN (or no greater than 2.5 times ULN if alkaline phosphatase no greater than ULN)
* Alkaline phosphatase no greater than ULN (or no greater than 5 times ULN if AST/ALT no greater than ULN)
* No history of chronic hepatitis

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No uncontrolled congestive heart failure
* No uncontrolled angina
* No myocardial infarction and/or stroke within the past 6 months
* No active thromboembolic event within the past 4 weeks

Gastrointestinal:

* No gastrointestinal bleeding within the past 6 months
* No history of peptic ulcer disease

Other:

* No prior hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No prior allergy to any non-steroidal anti-inflammatory drug
* No other prior or concurrent malignancy within the past 3 years except adequately treated squamous cell or basal cell skin cancer or carcinoma in situ of the cervix
* No grade 2 or greater peripheral neuropathy
* No other serious concurrent medical illness
* No history of dementia, active psychiatric disorder, or other condition that would interfere with ability to take oral medication or preclude compliance with study
* HIV negative
* Must weigh at least 50 kg (110 pounds)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior biologic therapy for NSCLC

Chemotherapy:

* No prior chemotherapy for NSCLC

Endocrine therapy:

* At least 3 days since prior steroids

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to target lesion

Surgery:

* At least 4 weeks since prior major surgery

Other:

* Prior intermittent use of non-steroidal anti-inflammatory drugs (NSAIDs), including rofecoxib or celecoxib, allowed
* At least 1 week since prior fluconazole
* No recent prior NSAIDs, including rofecoxib or celecoxib, for a duration of more than 30 consecutive days
* No concurrent fluconazole or lithium
* No concurrent NSAIDs except aspirin administered at a dose of no more than 325 mg/day for cardiovascular conditions
* No other concurrent cyclo-oxygenase-2 inhibitors
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2001-10; Primary Completion 2005-09 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of combining celecoxib with docetaxel in elderly (> or = 70 yrs old) or poor performance status (PS)of 2 | Weeks 1, 2, and 3
  Blood levels of VEGF & PGE2

SECONDARY OUTCOMES:
Response rate of Celecoxib and Docetaxel | Every 2 cycles (or every 42 days); After therapy is completed or if the patient is only on Celecosxib, will be assessed for progression every month by clinical exam and every 3 months by radiological evaluation.
  CT Chest/Abdomen
Toxicity of Celecoxib and Docetaxel | Weeks 1, 2, and 3 of each 28 day cycle
  Routine bloodwork
Expression of cyclooxygenase-2 (COX-2) in tumors | Pre-Study
  Tissue sample from initial diagnosis, parrafin embedded tissue block
Changes in plasma levels of prostaglandin E2(PGE2) & vascular endothelial growth factor (VEGF) | Pre-study, Weeks 1, 2 and 5
  Collecting blood plasma

CONTACTS AND LOCATIONS:
Overall Officials: Shirish M. Gadgeel, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- [Result] Gadgeel SM, Wozniak A, Ruckdeschel JC, Heilbrun LK, Venkatramanamoorthy R, Chaplen RA, Kraut MJ, Kalemkerian GP. Phase II study of docetaxel and celecoxib, a cyclooxygenase-2 inhibitor, in elderly or poor performance status (PS2) patients with advanced non-small cell lung cancer. J Thorac Oncol. 2008 Nov;3(11):1293-300. doi: 10.1097/JTO.0b013e31818b194e. PMID 18978565
- [Result] Gadgeel SM, Shehadeh N, Kraut MJ, et al.: Preliminary results of a phase II study of celecoxib and weekly docetaxel in elderly (>70 yrs) or PS2 patients with advanced non-small cell lung cancer (NSCLC). [Abstract] Lung Cancer 41 (Suppl 2): A-O-110, S35, 2003.